CLINICAL TRIAL: NCT00874900
Title: Asthma Learning Project: Randomized Trial of a Computerized Asthma Game in a Pediatric Emergency Department
Brief Title: Asthma Learning Project
Acronym: ALP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Julie Brown, MD, MPH, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALP12526
Record Dates: First submitted 2009-04-01; First posted 2009-04-03 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2011-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Game (Experimental)
  Interventions: Other: Educational game
- Game + Activation (Experimental)
  Interventions: Other: Educational game + motivational interview
- Booklet (No Intervention)
- Booklet + Activation (Experimental)
  Interventions: Other: Motivational interview

INTERVENTIONS:
Other: Educational game — "Quest for the Code" is an educational asthma computer game. Participants randomized to this intervention will have access to the game for a minimum of one hour while receiving treatment in the Seattle Children's Emergency Department.
  Arms: Game
Other: Educational game + motivational interview — "Quest for the Code" is an educational asthma computer game. Participants randomized to this intervention will have access to this game for a minimum of one hour while receiving treatment in the Seattle Children's Emergency Department (ED).Before leaving the ED, participants in this group will have a brief asthma goal setting activity using motivational interview techniques.
  Arms: Game + Activation
Other: Motivational interview — Participant randomized to this group will receive standard care for the treatment of their asthma, including an education asthma booklet developed by Seattle Children's. Before leaving the ED, participants in this group will have a brief asthma goal setting activity using motivational interview techniques.
  Arms: Booklet + Activation

SUMMARY:
The purpose of this study is to determine the effect on knowledge and behavior of playing an educational asthma computer game during a pediatric Emergency Department (ED) asthma visit among children ages 7 - 15 years. The ED cares for a high-risk population of children who have difficulty accessing preventive care well. The addition of a computer game to usual asthma emergency care could be a simple, effective, enjoyable way to improve patients' asthma knowledge, beliefs, and management practices. This project has the potential to lead to larger studies evaluating the benefit of education with and without behavioral interventions such as motivational interviewing.

This project plans to implement and evaluate the use of a goal setting activity and the educational asthma computer game, "Quest for the Code" (Starlight Starbright Children's FoundationTM), in the ED of Seattle Children's Hospital. In a randomized trial of Spanish and English speaking children ages 7 - 15 years receiving ED care for their asthma, the investigators will evaluate the effects of the game on children's asthma knowledge, attitudes, and behaviors.

The investigators aim to compare the change in asthma knowledge and locus of control after 3 months, for children who play the computerized asthma game, versus those who receive standard care in the ED. The investigators will also compare changes in asthma severity and activity limitations over 3 months, for children who play the asthma game without goal-setting, children who playing the game with goal-setting, and children who receive standard care.

Overall, the investigators hypothesize that educational asthma game play by pediatric patients with acute asthma will improve asthma knowledge, compared with standard care.

ELIGIBILITY:
Inclusion Criteria:

* Age 7 - 15 years, inclusive.
* Patient has a history of asthma or asthma-like symptoms on at least 1 occasion, occurring at least 3 months prior to the current episode (may be verbal per patient/caregiver).
* Patient is presenting to the ED for an acute asthma exacerbation of any type or severity.
* Available for phone call or mail questionnaire in 2 weeks and 3 months.
* Parent able to read English or Spanish.
* Child able to understand spoken English or Spanish.
* Child able to use a computer and mouse or stylus.
* Provider believes the patient is likely to remain in ED for at least one hour.
* Informed consent by parent and assent from child

Exclusion Criteria:

* Child has previously participated in this study.
* Child has a hearing impairment uncompensated for by assistive listening devices.
* Significant mental disorder or cognitive impairment that the parent believes would preclude competent informed assent or game play.
* Child has a baseline motor disorder and the parent is unable to assist using a mouse and keyboard
* Child has significant medial conditions that have a pulmonary component, in addition to their asthma

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2008-12; Primary Completion 2013-01 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Child Knowledge | 3 months

SECONDARY OUTCOMES:
Locus of control | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Julie Brown, MD, MPH, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States